CLINICAL TRIAL: NCT02757183
Title: Do Patient-Centric mHealth Programs Improve Patient Engagement and Health Outcomes.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: AnalyticsPlus, Inc. (Industry)
Collaborators: Cedars-Sinai Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: Pro-00041208-AP
Record Dates: First submitted 2016-04-27; First posted 2016-05-02 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: "IntelliH" — "IntelliH" is a mobile health and a web-based software application that allows patients to enter their blood glucose, weight, medication, diet and other life-style data for review by their providers and monitor their health remotely.

SUMMARY:
The "INTELLIH" (brand name of the mobile health application) Diabetes Study is to understand the usage of a mobile health application, IntelliH, and connected wireless devices such as glucometer by the diabetic patients and ascertain if there are any improvements in short-term health outcomes.

DETAILED DESCRIPTION:
The proposed pilot program is the first of its kind in the nation to use a product, "IntelliH" - Intelligent Health for All, that combines four key technologies in one platform: 1) Mobile health application (mHealth) App and web portal, 2) wireless sensors and wearable devices, 3) Secure text messaging when both sender and receiver are logged in to the system and video-based patient interaction, and 4) remote health monitoring. The purpose of this pilot program is to understand a) usage and adoption of these technologies by providers and patients, and b) document the short-term improvements in health outcomes in a diabetic population. This pilot study will follow 20 diabetic patients (Type 1 or Type 2) as they beta-test this system, and will acquire data on consented subjects over a period of six months.

ELIGIBILITY:
Inclusion Criteria:

* A1c greater than or equal to 6.5%.
* Age greater than or equal to 18 years.
* Ability to comply with study protocol.
* Available and usable internet facilities at home.
* Availability and usable smart phone.

Exclusion Criteria:

-Inability to comply with instructions and directions.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study participants will be recruited from the list of diabetes patients coming to Cedars-Sinai Medical Center for their regular treatment. Several physicians will be involved in making this program available to their patients. Eligible and consenting patients will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2016-04; Primary Completion 2016-11 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Usage and Adoption of the smart phone based mobile health application | Six Months
  Patients adoption will be assessed directly through the application and through questionnaire

SECONDARY OUTCOMES:
Blood glucose range maintenance and variation | Six months
  Frequency of hypoglycemic, hyperglycemic, and out of recommended range events
Adherence to Prescribed Medication | Six months
  Medication adherence rates will be measured for each medication used by patient

CONTACTS AND LOCATIONS:
Overall Officials: Ruchi Mathur, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided